## CONSENT DOCUMENT FOR PARTICIPATION IN A RESEARCH STUDY

TITLE: Comparative analysis of the effectiveness and safety of the Erectus Spinae Lumbar Plane

| block (ESP-L) versus no locoregional blo | ck in hip surgery |
|---|---|
| I | |
| • I read the above mentioned study part to chat withstudy. | ticipant information sheet that was given to me, I was able and ask all necessary questions about the |
| • I understand that my participation is time, without having to give explanations | voluntary, and that I can withdraw from the study at any and without this affecting my medical care. the conditions detailed in the participant information sheet. in this study. |
| Signed.: The participant, | Signed.: The researcher requesting consent |
| First and last name:<br>Date: | First and last name:<br>Date: |

## **DOCUMENT OF CONSENT BEFORE WITNESSES FOR PARTICIPATION IN A RESEARCH STUDY** (for cases where the participant cannot read/write)

The impartial witness will have to identify himself and be a person outside the investigative team

| TITLE Comparative analysis of th block (ESP-L) versus no locoregion | he effectiveness and safety of the Erectus Spinae Lumbar Plane<br>hal block in hip surgery |
|---|---|
| I | , as an impartial witness, affirm that in my |
| presence: | |
| • | has read the Participant Information Shee |
| <ul> <li>You understand that your partic<br/>any time, without having to give ex</li> </ul> | ven to you, and has been able to ask all questions about the study sipation is voluntary, and that you can withdraw from the study at planations and without this affecting your medical care. data under the conditions detailed in the information sheet for the participate in this study. |
| Signed.: The witness | Signed.: The researcher requesting consent |
| First and last name: Date: | First and last name: Date: |